CLINICAL TRIAL: NCT04380246
Title: COA-APTIC CLINICIAN CONCEPT ELICITATION STUDY: A Qualitative Concept Elicitation Study to Identify Important Aspects of Pain Assessment, Treatment, and Response to Treatment in Children Who Are 0 to <3 Years of Age
Brief Title: COA-APTIC Clinician Concept Elicitation Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00105109
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2020-04

CONDITIONS: Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinicians: Clinicians who care for pediatric patients >50% of their time, who treat pediatric patients who are in acute pain and between 0 and 3 years of age. May include physicians, clinical pharmacists, nurse practitioners, physician assistants, and/or nurses.
  This cohort will complete a qualitative interview about pain and distress in infants and young children.
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Other: Qualitative Interview — There is no intervention as part of this study. Clinicians will participate in a qualitative interview.

SUMMARY:
This is a concept elicitation study to identify important aspects of acute pain assessment, treatment, and response to treatment in infants and young children, age 0 to 3 years old, from a clinician's perspective.

DETAILED DESCRIPTION:
The purpose of this study is to identify important endpoints and outcomes for use in pediatric trials of acute pain therapeutics in children who are 0 to <3 years of age from a clinician's perspective. To identify these endpoints and outcomes the investigators will conduct remote qualitative concept elicitation interviews with 27 clinicians who treat pediatric patients. These interviews will include verbal consent to participate, a demographics questionnaire, and a semi-structured interview which will last approximately one hour. Interview questions will address the participant's professional experience recognizing and managing pain in children between 0 and 3 years of age. Interviews will be audio recorded and transcribed with the participant's permission. Transcripts and notes will be coded and analyzed. This is a minimal risk study; the investigators are only using standard interview procedures and are not collecting any protected health information from participants. While the investigators do not believe that any information collected would jeopardize the personal or professional standing of participants, all information will be kept strictly confidential per Good Clinical Practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Is a practicing clinician in a clinical care environment
2. Cares for pediatric patients >50% of their time
3. Treats or works with pediatric patients who are between 0 and <3 years of age AND being treated for acute pain
4. Holds one of the following titles/positions

   1. Physician
   2. Clinical pharmacist (PharmD)
   3. Nurse practitioner
   4. Physician assistant
   5. Nurse (with a BSN/RN or higher)
5. Is over the age of 18 years
6. Can speak and understand English
7. Is capable of giving informed verbal consent

Exclusion Criteria:

1. Lack of access to a telephone for interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be practicing clinicians who care for pediatric patients > 50% of their time, and who treat pediatric patients who are in acute pain and between 0 and 3 years of age
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Clinician perspectives on how to identify or recognize pain in children 0 to <3 years of age | 1 hour
  A 1-hour qualitative interview will be conducted and transcript or interviewer notes coded to assess how clinicians identify and recognize acute pain in infants and young children
Clinician perspectives on how and when to treat acute pain in children 0 to <3 years of age | 1 hour
  A 1-hour qualitative interview will be conducted and transcript or interviewer notes coded to assess how clinicians treat acute pain in infants and young children
Clinician perspectives on how to evaluate response to treatment for acute pain in children 0 to <3 years of age | 1 hour
  A 1-hour qualitative interview will be conducted and transcript or interviewer notes coded to assess how clinicians evaluate response to treatment for acute pain in infants and young children
Clinician perspectives on important side effects of acute pain therapeutics in children 0 to <3 years of age | 1 hour
  A 1-hour qualitative interview will be conducted and transcript or interviewer notes coded to assess important side effects of acute pain therapeutics in infants and young children

CONTACTS AND LOCATIONS:
Overall Officials: Bryce Reeve, PhD, Principal Investigator — Duke University; Kanecia Zimmerman, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of the study team.